CLINICAL TRIAL: NCT01280032
Title: Kypho-IORT: Phase II Study for Dose Escalation of Intraoperative Radiotherapy During Kyphoplasty for Spinal Metastases
Brief Title: Kypho-IORT: Intraoperative Radiotherapy During Kyphoplasty for Spinal Metastases
Acronym: Kypho-IORT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Frederik Wenz, Prof. Dr. med., Universitätsmedizin Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-Kypho-IORT-01
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Tumors
Keywords: intraoperative radiotherapy; kyphoplasty; spinal metastases
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kypho-IORT (Experimental)
  Interventions: Radiation: intraoperative radiotherapy

INTERVENTIONS:
Radiation: intraoperative radiotherapy — intraoperative radiotherapy (8 Gy) during kyphoplasty for spinal metatsases

SUMMARY:
Vertebral column is the most prevalent location of bone metastases. Besides axial pain, vertebral metastases cause pathological fracture and neurological dysfunction by spinal cord compression. Although the median overall survival of patients with bone metastases is only 7-9 month, half of them live longer and will require palliative treatment for their symptoms.

Treatment options are radiotherapy and /or surgical treatment such as laminectomy, vertebroplasty or kyphoplasty. Various studies have shown the superiority of postoperative external beam radiotherapy after kyphoplasty in spinal metastases compared to surgery or radiotherapy alone. Nevertheless postoperative radiation schedules last 2-4 weeks. Moreover many patients present visceral and bone metastases simultaneously and require urgent systemic therapy. However, due to potentiated toxicity, concurrent therapy with full dose chemotherapy and radiotherapy is rarely possible.

The investigators have therefore established a novel method for intraoperative radiotherapy (IORT) during kyphoplasty which enables immediate stability, sterilization of the metastasis and immediate initiation of chemotherapy.

The kyphoplasty itself is performed according to the standard procedure with some minor modifications. In short under general anaesthesia, a bipedicular approach into the affected vertebra is chosen with insertion of specially designed metallic sleeves to guide the electron drift tube of the miniature X-ray generator (INTRABEAM®). To perform the IORT during a kyphoplasty with this device a new applicator was designed. This sterile applicator consists of a plastic head, which is needed to attach it to the X-ray source and a stainless steel tube. This tube protects the probe from bending. Under fluoroscopic guidance the applicator including the drift tube is guided through the metallic sleeves in the vertebral body. A dose of 8 Gy in 5 mm distance is delivered. After IORT the INTRABEAM system is removed. The kyphoplasty balloon is inflated and PMMA-cement is injected. Afterwards the sleeves are removed and the wound is closed as usual.

Aim of this study is the definition of the maximum tolerable dose (MTD) for IORT during a kyphoplasty using specific MTD-criteria and evaluating the effectiveness of this combined treatment procedure. To determine the MTD 3 levels with increasing doses are planned:

8 Gy in 5 mm distance, 8 Gy in 8 mm distance and 8 Gy in 10 mm distance.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years
* Karnofsky Index ≥ 60
* histological or by imaging proven spinal metastases (2 cm diameter as the upper limit) inferior TH 3, which are accessible for kyphoplasty
* written informed consent obtained
* use of adequate contraceptive method by female patients of reproductive potential to minimize risk of pregnancy

Exclusion Criteria:

* uncontrolled intercurrent medical disorder - including but not limited to ongoing or active infection (including infections in the area of the treated spinal segment, for example, spondylitis / osteomyelitis / skin infections) or mental illness / social situation which affect the compliance of study requirements
* prior radiation of the same vertebra
* patients could not receive anaesthesia or surgery for medical reasons
* history of coagulation disorder associated with bleeding
* existing contraindications for MRI- or CT-scans
* pregnant or breast-feeding women

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
side effect of IORT using defined MTD criteria: dysfunction of wound healing, infections, osteoradionecrosis, nerve and spinal cord damage, pathological fracture within 90 days | 5 years

SECONDARY OUTCOMES:
Efficacy defined by CT or MR-imaging and / or clinical relapses / progress and pain | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiotherapy University Hospital Mannheim, Mannheim, Germany

REFERENCES:
- [Result] Bludau F, Winter L, Welzel G, Obertacke U, Schneider F, Wenz F, Ruder AM, Giordano FA. Long-term outcome after combined kyphoplasty and intraoperative radiotherapy (Kypho-IORT) for vertebral tumors. Radiat Oncol. 2020 Nov 12;15(1):263. doi: 10.1186/s13014-020-01715-z. PMID 33183307
- [Result] Bludau F, Welzel G, Reis T, Schneider F, Sperk E, Neumaier C, Ehmann M, Clausen S, Obertacke U, Wenz F, Giordano FA. Phase I/II trial of combined kyphoplasty and intraoperative radiotherapy in spinal metastases. Spine J. 2018 May;18(5):776-781. doi: 10.1016/j.spinee.2017.09.011. Epub 2017 Sep 28. PMID 28962909